CLINICAL TRIAL: NCT06072287
Title: Testing the Reliability and Validity of a New Measure for Illness-related Distress.
Brief Title: The Living With a Long-Term Condition Study
Acronym: LTC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: HR/DP-22/23-36320
Record Dates: First submitted 2023-10-02; First posted 2023-10-10 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-09

CONDITIONS: Asthma; Atrial Fibrillation; Cancer; Cerebrovascular Disorders; Stroke; CKD; Copd; Fibromyalgia; Pain; Heart Diseases; Heart Disease Chronic; Dementia; Diabetes; Epilepsy; Heart Failure; High Blood Pressure; Hypertension; Hiv; AIDS; IBD; IBS; Liver Diseases; Long COVID; Lupus Erythematosus; Multiple Sclerosis; Obesity; Osteoarthritis; Arthritis; Rheumatoid Arthritis; Osteoporosis; Parkinson Disease; Sickle Cell Disease; Hepatitis; Endometriosis; PCOS; Neurological Disorder; POTS - Postural Orthostatic Tachycardia Syndrome; MND (Motor Neurone DIsease); Cystic Fibrosis; Migraine; Spondylitis; Celiac Disease; Hidradenitis Suppurativa; Eczema; ME/CFS
Keywords: mental health; depression; anxiety; chronic illness
MeSH Terms: conditions — Asthma; Atrial Fibrillation; Neoplasms; Cerebrovascular Disorders; Stroke; Pulmonary Disease, Chronic Obstructive; Fibromyalgia; Pain; Heart Diseases; Dementia; Diabetes Mellitus; Epilepsy; Heart Failure; Hypertension; Acquired Immunodeficiency Syndrome; Liver Diseases; Post-Acute COVID-19 Syndrome; Multiple Sclerosis; Obesity; Osteoarthritis; Arthritis; Arthritis, Rheumatoid; Osteoporosis; Parkinson Disease; Anemia, Sickle Cell; Hepatitis; Endometriosis; Nervous System Diseases; Postural Orthostatic Tachycardia Syndrome; Amyotrophic Lateral Sclerosis; Cystic Fibrosis; Migraine Disorders; Spondylitis; Celiac Disease; Hidradenitis Suppurativa; Eczema; Fatigue Syndrome, Chronic; Psychological Well-Being; Depression; Anxiety Disorders; Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Participants will answer two short questionnaires, 1 week apart.
  Interventions: Diagnostic Test: Living with LTC Questionnaire

INTERVENTIONS:
Diagnostic Test: Living with LTC Questionnaire — A questionnaire that will ask about demographic information, mental wellbeing and distress related to chronic illness.

SUMMARY:
Psychological distress (anxiety and depression) is common in and experienced differently by people living with long-term health conditions (LTCs). Being able to measure whether psychological distress is related to living with a LTC would allow researchers and clinicians to provide interventions specifically tailored to the challenges of living with a LTC and therefore provide the most appropriate support for these patients. Such a measure would also be useful in research to identify the presence of illness-related distress in different patient groups. This project will therefore create a new measure of illness-related distress that has applications for both research and clinical practice. This will involve the psychometric validation of the new illness-related distress measure to test how valid and reliable the measure is.

The aim of the project is to provide initial validation of the Illness Related Distress Scale in a community sample, recruited through online platforms. The objective of the study is to gather initial validity and reliability data for the scale.

DETAILED DESCRIPTION:
Background: see brief summary

Project information:

This study will be conducted online with participants from the UK. A series of standardised questionnaires will be used alongside the new questionnaire.

Participants will be those who self-select to complete our survey by responding to advertisements. The invitation will include a link to the Qualtrics survey which includes the Participant Information Sheet, Eligibility Screening, Consent Form and Baseline Questionnaire.

After completing eligibility screening and consent, participants will complete the baseline questionnaire which will include brief demographics (highest education level, long-term condition diagnoses, ethnicity age and gender), the new measure we are testing (the Illness Related Distress Scale), as well as the Patient Health Questionnaire (PHQ-8), Generalised Anxiety Disorder Scale (GAD-7), the Work and Social Adjustment Scale (WSAS). The baseline questionnaire will only include the Inflammatory Bowel Disease Distress Scale (IBD-DS) and Diabetes Distress Scale (DDS) if participants indicate that they have a diagnosis of the relevant condition.

At 1 week follow-up, participants will be sent a Qualtrics link to complete our 1-week follow-up questionnaire which will include the new Illness-Related Distress Scale only.

Participants:

We are aiming to recruit 600-700 participants for the study.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Self-reported diagnosis of a Long-Term Condition
* UK resident
* Possession of an email address to enable all study procedures
* Sufficient command of written and spoken English to understand study procedures

Exclusion Criteria:

* Under the age of 18
* Not living in the UK
* No self-reported diagnosis of an LTC
* Inability to complete questionnaires in English

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults in the UK with a diagnosis of a Long-Term Condition or chronic illness.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-10 (Estimated)

PRIMARY OUTCOMES:
Illness-related distress | Week 0 and Week 1
  31 item questionnaire developed by the research team designed to assess illness-related distresss.

SECONDARY OUTCOMES:
Depression | Week 0
  Eight-item Patient Health Questionnaire - 8 (PHQ-8) Minimum=0, maximum=24, with higher scores indicating greater depression.
Anxiety | Week 0
  Seven-item Generalised Anxiety Disorder Scale (GAD-7). Minimum=0, maximum=21, with higher scores indicating greater anxiety.
Functional impairment | Week 0
  Five-item Work and Social Adjustment Scale (WSAS). Minimum=0, maximum=50, with higher scores indicating greater functional impairment.
Diabetes Related Distress Scale | Week 0
  Diabetes Related Distress Scale (DDS-17), a 17 item self-report diabetes related distress questionnaire. Minimum=17, maximum=102, with higher scores indicating greater distress.
IBD Distress Scale | Week 0
  IBD Distress Scale, a 28 item self-report IBD related distress questionnaire. Minimum=29, maximum=145, with higher scores indicating greater distress.
Cognitive and Behavioural Responses to Symptoms | Week 0
  Cognitive Behavioural Responses to Symptoms Questionnaire, 40 item self-report questionnaire consisting of seven subscales with items scored on a 5 point scale. Higher scores correspond with stronger presence of the specific cognitive/behavioural response. The seven subscales refer to 1) fear avoidance, 2) catastrophising, 3) damage beliefs, 4) embarassment avoidance 5) symptom focussing 6) all-or-nothing behaviour and 7) avoidance/resting behaviour.

CONTACTS AND LOCATIONS:
Overall Officials: Rona Moss-Morris, PhD, Principal Investigator — King's College London; Annie Jones, PhD, Study Director — King's College London; Emma Jenkinson, MSc, Study Director — King's College London; Natasha Seaton, MSc, Study Director — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Study information and sign up — https://linktr.ee/ltc_study